CLINICAL TRIAL: NCT00698386
Title: Efficacy of Oral Zinc Administration as an Adjunct Therapy in Category I Pulmonary Tuberculosis Along With Assessment of Immunological Parameters (Double-blind, Randomized, Placebo-Controlled, Multicenter Clinical Trial
Brief Title: Efficacy of Oral Zinc Administration as an Adjunct Therapy in New Pulmonary Tuberculosis (Category I) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology, India (Other Government)
Responsible Party: Surendra Kumar Sharma, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTPR7885/Med/141166/06
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2008-06

CONDITIONS: Pulmonary Tuberculosis
Keywords: Micronutrient Zinc; Category I PTB; RNTCP; DOTS; Sputum smear conversion; Reduced relapse; Immunopathogenesis; Category-I
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Zinc supplement — Zinc miconutrient supplements have been prepared by Cadila pharmaceutical Ltd., India, in the form of capsules.Each micronutrient capsule contains 50mg zinc (as zinc sulphate) in a lactose matrix.In this clinical trial one tablet of zinc as oral supplement will be given everyday during the entire course in line with the directly observed treatment, short-course (DOTS) strategy recommended by the World Health Organization.
Dietary Supplement: Placebo — Placebo have been prepared by Cadila pharmaceutical Ltd., India, in the form of capsules.The placebo consisted of lactose alone. Supplement and placebo capsules were indistinguishable in appearance both externally and internally.

SUMMARY:
The primary objective of the study is to evaluate the efficacy of oral Zinc administration in new smear positive pulmonary tuberculosis patients. Evidence is available suggesting that zinc deficiency rapidly diminishes antibody- and cell-mediated immune responses in both humans and animals and renders the individual susceptible to a variety of pathogens. This micronutrient has also been found to be useful in the treatment of lung tuberculosis in limited number of patients.

We are conducting this study in category-I patients (As per World Health Organization, Geneva classification of tuberculosis) having lung tuberculosis to see the efficacy and also to see any change in the immunological parameters.

DETAILED DESCRIPTION:
Malnutrition is commonly observed in patients with pulmonary tuberculosis. There are reports claiming patients with active pulmonary tuberculosis are malnourished as indicated by diminished visceral proteins, anthropometric indexes, and micronutrient status. Zinc plays role in protecting cells from the damaging effects of free radicals. Zinc supplementation was shown to prevent pulmonary pathology due to hypoxia-induced lung damage in rats. The role of zinc in faster sputum smear conversion has not yet been studied. However, there are reports which confirms, in vitro cellular killing of tubercle bacilli by macrophages after zinc supplementation.

We are investigating oral zinc supplement for its efficacy in TB patients in a "double-blind placebo-controlled randomized clinical trial" fashion. We are conducting this trial in Category-I pulmonary TB Patients (as per RNTCP, Ministry of Health and Family Welfare, Govt.of India), and are assessing the outcome in the form of clinical improvement, sputum conversion and immunological parameters. This is a multi-centric trial sponsored by the Department of Biotechnology, Ministry of Science and Technology, Govt. of India.

Supplements and placebo have been prepared by Cadila pharmaceutical Ltd., India, in the form of tablets. Each micronutrient tablet contains 50mg zinc (as zinc sulphate) in a lactose matrix. The placebo consisted of lactose alone. Supplement and placebo capsules were indistinguishable in appearance both externally and internally. In this clinical trial one tablet of zinc as oral supplement will be given everyday during the entire course in line with the directly observed treatment, short-course (DOTS) strategy recommended by the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed sputum smear positive pulmonary TB cases.

Exclusion Criteria:

* Hypersensitivity to Category I anti-TB drugs.
* Category II pulmonary TB and multi-drug resistant TB (MDR-TB). patients.
* Presence of secondary immunodeficiency states: HIV, organ transplantation, diabetes mellitus, malignancy, treatment with corticosteroids Hepatitis B and C positivity.
* Patients with extrapulmonary TB and/or patients requiring surgical intervention.
* Currently receiving cytotoxic therapy, or have received it within the last 3 months.
* Pregnancy and lactation.
* Patients with a known seizure disorder.
* Patients with known symptomatic cardiac diseases, such as arrhythmias or coronary artery disease.
* Patients with abnormal renal function (serum creatinine more than 2 mg/dl or more than 2+ proteinuria or both).
* Patients with abnormal hepatic functions (serum bilirubin > 1.5 mg/dl; AST, ALT, SAP more than 1.5 times of upper limit of normal; PT = 1.3 times of control).
* Patients with hematological abnormalities (WBC lesser than or equal to3000/ cubic mm; platelets less than or equal to 100,000/cubic mm).
* Seriously ill and moribund patients with complications: low lung reserve, marked tachypnoea, chronic corpulmonale, congestive cardiac failure, BMI<15, severe hypoalbuminemia.
* Patients unable to survive for less than 6 months.
* Patients unable to comply with the treatment regimen.
* Patients with history of alcohol or drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The time of sputum conversion as well as the early sputum conversion from the baseline between the two groups will be evaluated. | 6 months
The cure rate will be evaluated as the primary parameter of efficacy. | 6 months
The relapse at an interval of 6,12,18 and 24 months after the completion of the therapy in patients of category-I pulmonary TB will be compared in both the groups. | 30 months
Recording of any clinical adverse reactions at anytime during the study for assessment of safety. | 30 months

SECONDARY OUTCOMES:
An additional secondary efficacy endpoint is the patient's and physician's global assessment of the clinical cure. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra Kumar Sharma, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medcial Sciences-, New Delhi, New Delhi, India